CLINICAL TRIAL: NCT06463301
Title: Effects of Treadmill Training on Motor Function, Balance, and Spasticity Reduction in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RIPHAH/FR&AHS-01827
Record Dates: First submitted 2024-04-29; First posted 2024-06-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Training in cp child (Experimental): Treadmill training for children should be carefully tailored to their developmental level, physical ability, and specific therapeutic goals. Initial Sessions start with shorter sessions, around 5-10 minutes, especially for children with disabilities.
  Progression will be made when the child becomes more accustomed to the treadmill. Aim for a total of 20-30 minutes per session, including breaks if necessary then then Start at a slow walking pace, approximately 0.5 to 1.0 miles per hour (mph) or 0.8 to 1.6 kilometers per hour (kph). Adjust the speed based on the child's comfort and ability to maintain a safe and effective walking pattern.
  Older Children (8-12 years Begin with a walking pace of 1.0 to 1.5 mph (1.6 to 2.4 kph). Gradually increase the speed to a brisk walk or light jog, up to 2.0 to 3.0 mph (3.2 to 4.8 kph), depending on the child's progress and comfort level along with conventional physical therapy
  Interventions: Other: Treadmill Training In CP child
- Conventional Physical therapy (Active Comparator): conventional physical therapy session would typically include gentle stretching, joint mobilization, range of motion exercises for both the upper and lower body, gait training, and standing frame activities. Each component is designed to improve various aspects of physical function, ensuring a comprehensive approach to rehabilitation
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Treadmill Training In CP child — Treadmill training for children should be carefully tailored to their developmental level, physical ability, and specific therapeutic goals. Initial Sessions start with shorter sessions, around 5-10 minutes, especially for children with disabilities.
  Progression will be made when the child becomes more accustomed to the treadmill. Aim for a total of 20-30 minutes per session, including breaks if necessary then then Start at a slow walking pace, approximately 0.5 to 1.0 miles per hour (mph) or 0.8 to 1.6 kilometers per hour (kph). Adjust the speed based on the child's comfort and ability to maintain a safe and effective walking pattern.
  Older Children (8-12 years Begin with a walking pace of 1.0 to 1.5 mph (1.6 to 2.4 kph). Gradually increase the speed to a brisk walk or light jog, up to 2.0 to 3.0 mph (3.2 to 4.8 kph), depending on the child's progress and comfort level along with conventional physical therapy.
  Arms: Treadmill Training in cp child
Other: Conventional Physical Therapy — conventional physical therapy session would typically include gentle stretching, joint mobilization, range of motion exercises for both the upper and lower body, gait training, and standing frame activities. Each component is designed to improve various aspects of physical function, ensuring a comprehensive approach to rehabilitation
  Arms: Conventional Physical therapy

SUMMARY:
This study investigates the impact of treadmill training on motor function, balance, and spasticity reduction in children with cerebral palsy (CP). The study synthesizes existing research to provide insights into the effectiveness of treadmill training as an intervention for improving these key outcomes in children with Cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy is a neurodevelopmental disorder characterized by impaired movement and posture due to non-progressive brain damage occurring before, during, or shortly after birth.this systematic review and meta-analysis comprehensively examines the effects of treadmill training on motor function, balance, and spasticity reduction in children diagnosed with cerebral palsy (CP).

The review includes studies published in peer-reviewed journals, databases, and relevant conference proceedings. Inclusion criteria encompass randomized controlled trials, quasi-experimental studies, and cohort studies evaluating treadmill training interventions in children aged 2-18 years with CP. Studies utilizing various treadmill training protocols, such as body-weight-supported treadmill training, overground treadmill training, or virtual reality-assisted treadmill training, are considered.

The primary outcomes assessed include changes in motor function, as measured by standardized assessment tools like the Gross Motor Function Measure (GMFM) or the Movement Assessment Battery for Children (MABC). Additionally, balance improvements are evaluated using validated balance assessment scales, while spasticity reduction is measured through clinical assessments, such as the Modified Ashworth Scale (MAS) or the Tardieu Scale.

The review aims to provide evidence-based insights into the efficacy of treadmill training as a rehabilitation intervention for children with CP, informing clinical practice guidelines and therapeutic decision-making. The findings contribute to our understanding of the potential benefits of treadmill training in improving motor function, balance, and spasticity in this

ELIGIBILITY:
Inclusion Criteria:

* Age 4 -12 years.
* Children having, I-II on GMFCM.
* Children diagnosed with spastic cerebral palsy.
* Children with will cognitive behavior

Exclusion Criteria:

* Misdiagnosed or not conform to Cerebral palsy.
* Children should be medically un stable uncontrolled seizures
* The children with mental retardation or other neurological disorders.
* Children with serve respiratory dysfunction, multiple contracture.
* Children with prior undone this type of training.
* Children with taking medication like muscle relaxant.
* Children having communication or hearing issues.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance scale to Measure balance | 12th weeks study , 1st reading will be take on baseline than after 4 weeks ,8weeks & 12weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (the lowest function) to 4 points (the highest function), with a maximum score of 56 points.in his study, we assessed the effect of treadmill training on balance of CP child

SECONDARY OUTCOMES:
Modified Ashworth Scale to measure spasticity | 12th weeks study , 1st reading will be take on baseline than after 4 weeks ,8weeks & 12weeks
  Ashworth Scale measures spasticity in patients with lesions to the central nervous system. AS is an assessment that is used to measure the increase in muscle tone. AS assigns a grade of spasticity from a 0-4 ordinal scale 0 means no spasticity 4 means complete rigidity
GMFCS (Gross Motor Function Classification System) to measure the motor functions | 12th weeks study ,1st reading will be take on baseline than after 4 weeks ,8weeks & 12weeks
  The GMFCS, or Gross Motor Function Classification System, is a five-level classification that differentiates children with cerebral palsy based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility.
  total score is 5 5 full dependent
  1 is independent of the limitation

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmad Awan, Phd, Principal Investigator — Riphah International University; Numan Sadiq, MS SPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Rehabilitation center, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grecco LA, Zanon N, Sampaio LM, Oliveira CS. A comparison of treadmill training and overground walking in ambulant children with cerebral palsy: randomized controlled clinical trial. Clin Rehabil. 2013 Aug;27(8):686-96. doi: 10.1177/0269215513476721. Epub 2013 Mar 15. PMID 23503736
- [Background] Chrysagis N, Skordilis EK, Stavrou N, Grammatopoulou E, Koutsouki D. The effect of treadmill training on gross motor function and walking speed in ambulatory adolescents with cerebral palsy: a randomized controlled trial. Am J Phys Med Rehabil. 2012 Sep;91(9):747-60. doi: 10.1097/PHM.0b013e3182643eba. PMID 22902937
- [Background] Mutlu A, Krosschell K, Spira DG. Treadmill training with partial body-weight support in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2009 Apr;51(4):268-75. doi: 10.1111/j.1469-8749.2008.03221.x. Epub 2009 Jan 21. PMID 19207302
- [Background] Mattern-Baxter K. Effects of partial body weight supported treadmill training on children with cerebral palsy. Pediatr Phys Ther. 2009 Spring;21(1):12-22. doi: 10.1097/PEP.0b013e318196ef42. PMID 19214072
- [Background] Mattern-Baxter K, Bellamy S, Mansoor JK. Effects of intensive locomotor treadmill training on young children with cerebral palsy. Pediatr Phys Ther. 2009 Winter;21(4):308-18. doi: 10.1097/PEP.0b013e3181bf53d9. PMID 19923970